CLINICAL TRIAL: NCT06457399
Title: The Effect of Heliox on the Work of Breathing in Adult Patients With Lower Airway Stenosis
Brief Title: Heliox on the Work of Breathing in Adult Patients With Lower Airway Stenosis
Status: Active, not recruiting | Type: Observational
Sponsor: Hospital Universitario 12 de Octubre (Other)
Responsible Party: Principal Investigator, Marta Corral Blanco, Principal Investigator, Hospital Universitario 12 de Octubre
Other Study IDs: HELIOX ON AIRWAY STENOSIS
Record Dates: First submitted 2024-05-30; First posted 2024-06-13 (Actual); Last update posted 2024-06-13 (Actual); Status verified 2024-06

CONDITIONS: Airway Obstruction
Keywords: Heliox; Airway Stenosis; Work of breathing; Airway resistance
MeSH Terms: conditions — Airway Obstruction | interventions — heliox; Oxygen

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Airway Stenosis: Patients with lower airway stenosis on waiting list for endoscopic intervention on stenosis by respiratory endoscopy unit.
  Interventions: Drug: Heliox; Drug: Oxygen

INTERVENTIONS:
Drug: Heliox — Treatment for 30 minutes with Heliox from a commercial tank (Oxhelⓒ, Air Liquideⓒ) with a fixed mixture of 70% helium and 30% oxygen with non-rebreather mask or reservoir bag at a flow of 12-15 lpm.
  Other Names: Helium - Oxygen
Drug: Oxygen — Treatment for 30 minutes with oxygen at FiO2 of 31% with Venturi mask.
  Other Names: Oxygen 31%

SUMMARY:
Heliox (a mixture of Helium and Oxygen) can reduce the work of breathing in patients with airway stenosis by modifying turbulent flow into laminar flow. The aim of this study was to analyze the effect of Heliox versus conventional oxygen therapy in patients with lower airway stenosis on muscular effort measured by electromyography and diaphragmatic ultrasound, thoracoabdominal synchrony assessed with plethysmographic bands, dyspnea, stridor, oxygen saturation, transcutaneous carbon dioxide value, blood pressure, heart rate and respiratory rate.

DETAILED DESCRIPTION:
Lower airway stenosis results in increased work of breathing with stridor and dyspnea, as a consequence of the increased resistances caused by the reduction in airway diameter. Airway resistance also depends on the length of the airway and the type of gas flow. Heliox (a mixture of Helium and Oxygen) is a gas less dense than air, which can change the flow from turbulent to laminar, reducing airway resistance by 20 to 40%, and therefore decreasing the work of breathing. Heliox is an inert gas that does not react with biological membranes, so there are few complications associated with its use, the most relevant being hypoxemia when fixed mixtures are not used and the the fraction of inspired oxygen (FiO2) supplied is less than 21%. The aim of the study was to evaluate if during the perioperative period of lower airway stenosis the administration of Heliox compared to oxygen could reduce the work of breathing and improve dyspnea. For this purpose, patients were treated for 30 minutes with Heliox (fixed mixture of 70% helium and 30% oxygen) using a non rebreather mask or reservoir bag versus 30 minutes with oxygen 31% using a Venturi mask.

ELIGIBILITY:
Inclusion Criteria:

* Patients with lower airway stenosis evaluated at the Respiratory Endoscopy Unit of the Hospital Universitario 12 de Octubre on the waiting list for endoscopic intervention on stenosis.
* Stenosis grade ≥ 3 and Borg scale score > 2.

Exclusion Criteria:

* Presence of relevant comorbidities (uncontrolled ischemic heart disease, ventricular dysfunction, pneumopathies with severe respiratory insufficiency, severe pulmonary hypertension).
* Inability to perform the test due to severe dyspnea or need for emergency intervention.
* Patient on continuous mechanical ventilation, invasive or non-invasive.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients will be recluted from the pneumology outpatient clinic of the Hospital 12 de Octubre
Sampling Method: Non-Probability Sample
Enrollment: 18 (Actual)
Dates: Start 2022-04-27 (Actual); Primary Completion 2023-05-31 (Actual); Study Completion 2024-11 (Estimated)

PRIMARY OUTCOMES:
Changes in Neural Ventilatory Drive (%): | 30 minutes with Heliox and 30 minutes with Oxygen 31%
  Percentage over the Root Mean Square peak for parasternal electromyography (EMG): averaged of the square root of the peak value and the area under the curve of parasternal EMG (%RootMeanSquare) adjusted for respiratory frequency, as a surrogate of diaphragmatic EMG, and sternocleidomastoid EMG, which will give us information on accessory muscle activation.

SECONDARY OUTCOMES:
Diaphragmatic excursion assessed with ultrasound | At minute 15 during the Heliox test and at minute 15 during the Oxygen 31% test.
  Assessment of muscular effort by measuring the diaphragmatic excursion (mm) at tidal volume and at vital capacity.
Thickening fraction of the diaphragm assessed by ultrasound | At minute 15 during the Heliox test and at minute 15 during the Oxygen 31% test.
  Assessment of muscular effort by measuring the thickening fraction of the diaphragm in the apposition zone (%).
Changes in thoracoabdominal synchrony | Phase angle was calculated from 10 consecutive breaths at minutes 1, 5, 15 and 30 during the Heliox test and the Oxygen 31% test.
  Assessment of thoracoabdominal synchrony using thoracic and abdominal belts by calculating the phase angle with the Lissajoux loop method (plotting abdominal motion on the x-axis against thoracic motion on the y-axis).
Borg Scale Dyspnea evolution (points) | Basal value and at minutes 1, 5, 15 and 30 during the Heliox test and the Oxygen 31% test.
  Degree of dyspnea will be determined by this validated scale with a result between 1 and 10 points.0: Not at all 0.5: Very, very light (hardly noticeable) 1: Very light, 2: Light, 3: Moderate , 4: Somewhat intense, 5: Intense, 6: Between 5 and 7, 7: Very intense, 8: Between 7 and 9, 9: Very, very intense (almost maximum ), 10: Maximum
Oxygen saturation | Basal value and at minutes 1, 5, 15 and 30 during the Heliox test and the Oxygen 31% test.
  Measured by pulse-oximetry
Transcutaneous partial pressure of carbon dioxide | Basal value and at minutes 1, 5, 15 and 30 during the Heliox test and the Oxygen 31% test.
  Transcutaneous monitor uses a noninvasive technique to measure the skin-surface partial pressure of carbon dioxide (PtcCO2)
Blood pressure | Basal value and at minutes 1, 5, 15 and 30 during the Heliox test and the Oxygen 31% test.
  Non-invasive measurement with a sphygmomanometer
Heart rate | Basal value and at minutes 1, 5, 15 and 30 during the Heliox test and the Oxygen 31% test.
  number of beats per minute
Respiratory rate | Basal value and at minutes 1, 5, 15 and 30 during the Heliox test and the Oxygen 31% test.
  Number of breaths per minute

CONTACTS AND LOCATIONS:
Overall Officials: Marta Corral Blanco, MD, Principal Investigator — Hospital 12 de Octubre
Locations (1):
- Marta Corral Blanco, Madrid, Spain